CLINICAL TRIAL: NCT00004829
Title: Phase III Randomized Study of the Inhalation of Tobramycin in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13390; PATH-PG-TNDS-002/003; PATH-FDR001235
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-06

CONDITIONS: Cystic Fibrosis; Bacterial Infection
Keywords: bacterial infection; cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; immunologic disorders and infectious disorders; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Bacterial Infections; Respiratory Tract Diseases; Genetic Diseases, Inborn; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Tobramycin

INTERVENTIONS:
Drug: tobramycin

SUMMARY:
OBJECTIVES: I. Determine the safety and efficacy of tobramycin in patients with cystic fibrosis who are chronically colonized with Pseudomonas aeruginosa.

II. Determine whether this treatment produces tobramycin-resistant bacteria at a frequency different from the placebo group and whether the emergence of resistance is associated with a lack of clinical response.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study.

Patients receive tobramycin or placebo by inhalation twice daily for 28 days followed by 28 days of rest. This treatment is repeated twice, for a total of 3 courses of therapy.

Patients are followed every 2 weeks for the first 8 weeks, then every 4 weeks, and then at 4 weeks after the last treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Documented cystic fibrosis with Pseudomonas aeruginosa present in a sputum or throat culture within 6 months prior to screening

Sweat chloride at least 60 mEq/L

--Prior/Concurrent Therapy--

At least 14 days since prior intravenous or aerosolized tobramycin or other antipseudomonal antibiotic

At least 4 weeks since prior administration of any investigational drug

No concurrent antibiotics by aerosol

--Patient Characteristics--

Renal:

* Creatinine less than 2 mg/dL
* BUN less than 40 mg/dL
* No proteinuria of 2+ or greater

Pulmonary:

* FEV1 at least 75% and at least 25% of predicted
* Room air oximetry at least 88% saturation
* Able to perform pulmonary function tests
* No hemoptysis of 60 mL or greater within 30 days prior to study
* No abnormal chest X-ray

Other:

* Not pregnant
* Fertile females must use effective contraception
* No history of positive culture with Burkholderia cepacia
* No history of glucose-6-phosphate dehydrogenase deficiency
* No known local or systemic hypersensitivity to aminoglycosides, albuterol, or other beta-2 agonists

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1995-06; Study Completion 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bruce Montgomery, Study Chair — Pathogenesis

REFERENCES:
- [Background] Ramsey BW, Pepe MS, Quan JM, Otto KL, Montgomery AB, Williams-Warren J, Vasiljev-K M, Borowitz D, Bowman CM, Marshall BC, Marshall S, Smith AL. Intermittent administration of inhaled tobramycin in patients with cystic fibrosis. Cystic Fibrosis Inhaled Tobramycin Study Group. N Engl J Med. 1999 Jan 7;340(1):23-30. doi: 10.1056/NEJM199901073400104. PMID 9878641